CLINICAL TRIAL: NCT06115954
Title: The Efficacy of Telerehabilitation-Based Self-Management Supported Exercise in Children and Adolescents With Juvenile Idiopathic Arthritis: A Randomized Controlled Study
Brief Title: Self-Management Supported Telerehabilitation in Children and Adolescents With Juvenile Idiopathic Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Berna Cagla Balkisli, Msc. Lecturer, Specialist Physiotherapist, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PamukkaleUni.
Record Dates: First submitted 2022-12-16; First posted 2023-11-03 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Telerehabilitation; Juvenile Idiopathic Arthritis; Self-Management
MeSH Terms: conditions — Arthritis, Juvenile

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Synchronous Telerehabilitation (Experimental): On the basis of telerehabilitation, before starting both synchronous and asynchronous exercise therapy, a comprehensive self-management program will be provided.
  Self-management training will be shared online synchronously with the participants in this exercise group. The exercise program will consist of functional exercises focused on trunk stabilization, including warm-up and cool-down periods, 3 times a week for 12 weeks, and will be performed online by the physiotherapist. Exercise training will be completed with a 10-minute warm-up exercise followed by 40-minute trunk stabilization and functional exercises for the upper and lower extremities, followed by a 10-minute cooling-down program consisting of flexibility exercises. Progression in exercise training will be done by increasing the number of repetitions and adding elastic bands to the exercises.
  Interventions: Other: Self-Management Supported Telerehabilitation
- Asynchronous Telerehabilitation (Active Comparator): Self-management training will be delivered to the participants in this exercise group via video and they will be asked to watch it. The exercise program will consist of functional exercises focused on trunk stabilization, including warm-up and cool-down periods, 3 times a week for 12 weeks, and will be shared with the participants through videos taken by the physiotherapist. Exercise training will be completed with a 10-minute warm-up exercise followed by 40-minute trunk stabilization and functional exercises for the upper and lower extremities, followed by a 10-minute cooling-down program consisting of flexibility exercises. Participants will be checked weekly by phone to determine exercise tracking. Progression in exercise training will be achieved with new videos that include an increase in the number of repetitions of the participants and the addition of elastic bands to the exercises.
  Interventions: Other: Self-Management Supported Telerehabilitation

INTERVENTIONS:
Other: Self-Management Supported Telerehabilitation — Supporting the exercises with an internet-based environment and self-management training for Children and Adolescents with Juvenile Idiopathic Arthritis

SUMMARY:
Juvenile idiopathic arthritis (JIA) is the most common chronic rheumatic disease of unknown etiology in childhood. JIA covers several different subgroups and is predominantly manifested by peripheral arthritis. Joint swelling, effusion, tenderness, pain in JIA; causes functional limitations, fatigue and quality of life disorders. Chronic inflammation limits the patient's daily activities and productivity. Self-management is defined as an individual's ability to manage their symptoms, treatment, lifestyle changes, and the psychosocial and cultural consequences of health conditions. Good self-efficacy and coping skills reduce the health and financial burden on the individual as well as on health care, benefiting society in general. Telerehabilitation is the dissemination of rehabilitation services through communication technologies. In the literature, it is seen that the studies on internet-based exercise applications are limited. In the studies, people were encouraged to physical activity with an internet-based application and the benefits of being active were given within the scope of patient education, and it was reported that the level of physical activity effectively improved as a result. It can also increase endurance, has been reported to be safe and feasible. In our study, unlike the literature, the self-management program and exercise applications will be integrated into the internet-based telerehabilitation method, based on the fact that the exercise practices in JIA are effective in disease management and improvement of symptoms. Therefore, in our study; the effectiveness of telerehabilitation-based exercise methods to be applied additionally synchronously and asynchronously to self-management education in children and adolescents with JIA on pain, disease activity, functional status, fatigue, quality of life, psychosocial status, self-efficacy and satisfaction will be examined and compared.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with Juvenile Idiopathic Arthritis according to ILAR diagnostic criteria
* 8-18 years old
* Agreeing to do the exercises throughout the study
* Stable symptoms and medications
* Internet and computer access

Exclusion Criteria:

* Be younger than 8 years old
* Surgical or arthroscopic operation in the last 1 year
* Having any musculoskeletal disease or orthopedic, neurological, psychological disease that may prevent participation in exercise
* Presence of active synovitis and arthritis
* Active vestibular disease
* Family and patient's inability to adapt to the assessment
* Having a psychiatric illness that affects cooperation
* Having heart failure and lung pathology at a level that will affect activities of daily living

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 26 (Actual)
Dates: Start 2022-12-23 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Juvenile Idiopathic Arthritis Disease Activity Score (JADAS) | Change from baseline to three months
  It assess the disease activity in patients with JIA.
Childhood Health Assessment Scale (CHAQ) | Change from baseline to three months
  It assess the children's functional ability over the past week.
Pediatric Quality of Life Inventory (PedsQL) 3.0 Arthritis Module | Change from baseline to three months
  It assess the patient's quality of life in pediatric arthritis.
Pediatric Quality of Life Inventory Multidimensional Fatigue Scale (PedsQL-F) | Change from baseline to three months
  It assess the fatigue in children.

SECONDARY OUTCOMES:
Numeric Rating Scale | Change from baseline to three months
  It assess the pain.
5 times sit and stand test | Change from baseline to three months
  It assess the functional status, muscle strength an endurance.
6-Item Self-Efficacy Scale for Managing Chronic Diseases | Change from baseline to three months
  It assess the self-efficacy in patients with chronic diseases.
The Juvenile Arthritis Biopsychosocial and Clinical Questionnaire -JAB-Q | Change from baseline to three months
  It assess the biopsychosocial status in JIA patients.

CONTACTS AND LOCATIONS:
Overall Officials: Bilge Basakci Calik, Prof. Dr., Study Director — Pamukkale University
Locations (1):
- Pamukkale University School of Physical Therapy and Rehabilitation, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No